CLINICAL TRIAL: NCT03540992
Title: Development of Diagnostic and Treatment Strategy for Resistant Hypertension
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2017-1222
Record Dates: First submitted 2018-05-03; First posted 2018-05-30 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Resistant Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a registry study to examine the clinical features, blood pressure control rate, and clinical prognosis of resistant hypertension in Koreans. This study will register patients with resistance hypertension in eight tertiary hospitals in Korea and follow up them for three years. The prognosis will be analysed according to etiologies, achieved blood pressure, and types of antihypertensive medication.

DETAILED DESCRIPTION:
This study will enroll hypertensive patients who are in treatment or those who are referred from primary clinic based on inclusion or exclusion criteria. Basic clinical information, compliance with antihypertensive medications, concomitant use of other medications will be investigated and all patients will perform 24-hr ambulatory blood pressure measurement. Screening for renal artery stenosis and primary aldosteronism will be conducted. Office blood pressure will be taken every 3-6 months. Home blood pressure measurement and 24-hr ambulatory blood pressure measurement will be performed every year. The primary outcome is the newly developed MACE during the follow-up period. The secondary outcomes are newly developed target organ damage (LVH confirmed by echocardiography or EKG, carotid femoral PWV≥ 12m/s, microalbuminuria (Urine albumin-creatinine ratio ≥30 mg/g)) and decline of renal function (doubling of serum creatinine, dialysis). The follow-up period is 3 years.

ELIGIBILITY:
Inclusion Criteria:

1. 20 years and older
2. Office SBP>130 mmHg or office DBP >90 mmHg with 3 antihypertensive medications of different classes
3. Treated hypertensive patients with 4 antihypertensive medications of difference classes including diuretics

Exclusion Criteria:

1. desired life time under 6 months due to non-cardiovascular disease (e.g. cancer, sepsis)
2. women with pregnancy or on nursing
3. within the first three months after transplantation
4. acute renal allograft rejection
5. within six months after discharge from hospitalization for acute coronary syndrome (myocardial infarction, unstable angina) or acute stroke
6. systolic heart failure (LVEF ≤40%)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A pateint diagnosed with resistant hypertension
Sampling Method: Non-Probability Sample
Enrollment: 780 (Estimated)
Dates: Start 2018-02-14 (Actual); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiac events | 3 years
  Composite of cardiovascular death, myocardial infarction, stroke, admission for heart fails

SECONDARY OUTCOMES:
Progression of CKD | 3 years
  Start dialysis or doubling of serum creatinine
Target organ damages | 3 years
  Target organ damage: LVH confirmed by echocardiography or EKG; carotid femoral PWV≥ 12m/s; microalbuminuria (Urine albumin-creatinine ratio ≥30 mg/g)
Target blood pressure achievement | 3 years
  Target blood pressure: Achievement of BP below 130/80 or 140/90 mmHg

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology Severance Cardiovascular Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Lee CJ, Ha JH, Kim JY, Kim IC, Ryu SK, Rhee MY, Lee JH, Lee JH, Lee HY, Ihm SH, Chung JW, Choi JH, Shin J, Park S, Kario K. Office blood pressure threshold of 130/80 mmHg better predicts uncontrolled out-of-office blood pressure in apparent treatment-resistant hypertension. J Clin Hypertens (Greenwich). 2021 Mar;23(3):595-605. doi: 10.1111/jch.14113. Epub 2020 Dec 5. PMID 33280228